CLINICAL TRIAL: NCT02240784
Title: A Natural History Study of Acute Hepatic Porphyria (AHP) Patients With Recurrent Attacks
Brief Title: EXPLORE: A Natural History Study of Acute Hepatic Porphyria (AHP)
Status: Completed | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-AS1-NT-001
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Acute Hepatic Porphyria
Keywords: Porphyria; AIP; VP; HCP; Variegate; Coproporphyria
MeSH Terms: conditions — Coproporphyria, Hereditary; Porphyrias; Coproporphyria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and plasma samples for known proteins associated with porphyria attacks.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Hepatic Porphyria

SUMMARY:
The purpose of this study is to characterize the natural history and clinical management of Acute Hepatic Porphyria (AHP) patients with recurring attacks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged >/= 12 years
* Diagnosis of AHP [acute intermittent porphyria (AIP), variegate porphyria (VP), hereditary coproporphyria (HCP) and aminolevulinic acid dehydratase (ALAD) deficient porphyria (ADP)]
* Porphyria attacks in the past 12 months or receiving treatment to prevent attacks
* Willing to provide written informed consent, medical records, and to comply with study requirements

Exclusion Criteria:

• Current participation in a clinical trial of an investigational product

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute Hepatic Porphyria
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Medical history of AHP patients (Part A only) | Baseline to 6-Month Follow-Up Visit
Medication usage of AHP patients (Part A only) | Baseline to 6-Month Follow-Up Visit

SECONDARY OUTCOMES:
Plasma biomarkers (Part A only) | 0, 6 months and During Attacks
Porphyria signs and symptoms (Part A only) | 0, 2, 4, 6 months
Quality of Life (Part A only) | 0, 6 months
Urine biomarkers (Part A only) | 0, 6 months and During Attacks
Healthcare Utilization (Part A only) | 0, 6 months
Change in disease activity as measured by Quality of Life (Part B only) | 0, 6, 12, 18, 24, 30, 36 months
Change in disease activity as measured by Porphyria Screening/Follow Up Questionnaire (Part B only) | 0, 3, 6, 9, 12, 18, 24, 30, 36 months
Change in disease activity as measured by Brief Pain Inventory form (Part B only) | 0, 3, 6, 9, 12, 18, 24, 30, 36 months
Change in disease activity as measured by European Organization for Research and Treatment of Cancer (EORTC) Questionnaire (Part B only) | 0, 6, 12, 18, 24, 30, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (30):
- United States (8):
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Galveston, Texas
  - Clinical Trial Site, Salt Lake City, Utah
- Clinical Trial Site, Camperdown, New South Wales, Australia
- Clinical Trial Site, Leuven, Belgium
- Clinical Trial Site, Sofia, Bulgaria
- Clinical Trial Site, Prague, Czechia
- Clinical Trial Site, Helsinki, Finland
- Clinical Trial Site, Paris, France
- Clinical Trial Site, Chemnitz, Germany
- Clinical Trial Site, Petah Tikva, Israel
- Italy (2):
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Modena
- Clinical Trial Site, Mexico City, Mexico
- Clinical Trial Site, Rotterdam, Netherlands
- Clinical Trial Site, Bergen, Norway
- Clinical Trial Site, Warsaw, Poland
- Clinical Trial Site, Cape Town, South Africa
- Clinical Trial Site, Seoul, South Korea
- Spain (2):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Murcia
- Clinical Trial Site, Zurich, Switzerland
- Clinical Trial Site, Taipei, Taiwan
- United Kingdom (2):
  - Clinical Trial Site, Cardiff, Wales
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No